CLINICAL TRIAL: NCT01719120
Title: Internet-Based Self-Help Cognitive-Behavioral Therapy for Insomnia (CBTI): A Randomized Controlled Trial
Brief Title: Internet-Based Cognitive-Behavioral Therapy for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBTI-001
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive-Behavioral Therapy; Internet-Based; Self-Help; Randomized Controlled Trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Self-help CBT with tel. consultation (Experimental): Self-help CBT with tel. consultation (SHTC)group will receive telephone consultation provided by the investigator in addition to self-help cognitive-behavioral therapy once per week for 6 consecutive weeks.During the consultation, the investigator will answer questions about the treatment content, monitor whether the subjects read the assigned materials and comply with the tasks and procedures, and provide encouragement and support.
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Self-help CBT (Experimental): The subjects will receive self-help cognitive-behavioral therapy (SH)once per week for 6 consecutive weeks.
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Waiting-list control (WL) (No Intervention): Subjects in this group will not receive any kind of treatment during the waiting period. They will receive the treatment identical to the self-help group within 3 months from the baseline.

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — CBT for insomnia aims at changing dysfunctional cognitive beliefs and maladaptive behaviors contributed to the maintenance of insomnia. It involves 4 main components including behavioral, cognitive, educational, and relaxation treatments.
  Arms: Self-help CBT; Self-help CBT with tel. consultation

SUMMARY:
The aim of this study is to develop an Internet-based self-help therapy program for insomnia in Chinese language, and to conduct a randomized waiting-list controlled trial on the efficacy of Internet-based self-help therapy for insomnia.

DETAILED DESCRIPTION:
This study is a randomized controlled trial in patients with insomnia. Eligible subjects will be randomly assigned to self-help treatment with telephone consultation (SHTC), self-help treatment without telephone consultation (SH), or waiting-list control. The subjects will receive self-help treatment once per week for 6 consecutive weeks. In addition to self-help treatment, the subjects in SHTC group will receive telephone consultation once per week for 6 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged ≥18 years
* Predominant complaint of difficulty initiating or maintaining sleep or early morning awakening or nonrestorative sleep with associated distress or impairment in social, occupational and other important areas of functioning for at least 3 nights per week for at least 3 months based on self- administered questionnaire
* Able to read Chinese and type Chinese or English
* Have Internet access (PC/ mobile phone), and with an email address
* Willing to give informed consent and comply with the trial protocol

Exclusion Criteria:

* Have suicidal ideas based on self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sleep parameters (sleep onset latency, sleep efficiency, total sleep time, times of wakening during sleep) changes from baseline to 5-week posttreatment by subjective measures using sleep log. | Baseline, 1-week, 5-week, and 12-week posttreatment.
  12-week posttreatment is only for within-group comparison in treatment groups

SECONDARY OUTCOMES:
Self-rated sleep quality score measured by the Pittsburgh Sleep Quality Index (PSQI) questionnaire | Baseline, 1-week, 5-week, and 12-week posttreatment.
  12-week posttreatment is only for within-group comparison in treatment groups
Self-rated sleep-related cognition score measured by Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) | Baseline, 1-week, 5-week, and 12-week posttreatment.
  12-week posttreatment is only for within-group comparison in treatment groups
Self-rated severity of depressive and anxiety symptoms measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, 1-week, 5-week, and 12-week posttreatment
  12-week posttreatment is only for within-group comparison in treatment groups
Subjects' general health and quality of life regarding physical functioning, social functioning, physical role limitations, emotional role limitations, mental health, vitality, bodily pain, and general health perception measured by Short form -36 (SF-36) | Baseline, 1-week, 5-week, and 12-week posttreatment.
  12-week posttreatment is only for within-group comparison in treatment groups
Self-rated fatigue score measured by Multidimensional Fatigue Inventory (MFI) | Baseline, 1-week, 5-week, and 12-week posttreatment.
  12-week posttreatment is only for within-group comparison in treatment groups
Subjects' acceptability and credibility to the treatment measured by Treatment acceptability and credibility rating scale | Baseline and 1-week posttreatment
Subjects' adherence to the treatment measured by Treatment adherence rating scale | 1-week posttreatment
Subjects' satisfaction to the treatment measured by Treatment satisfaction rating scale | Treatment Week 2-6
Potential side effects associated with each component of CBT measured by Symptom checklist | Treatment Week 2-6 and 1-week posttreatment
Self-rated sleep quality score changes from baseline to 12-week posttreatment measured by Insomnia Severity Index questionnaire | Baseline, treatment Week 3, 1-week, 5-week and 12 week posttreatment.
  12-week posttreatment is only for within-group comparison in treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Fai Chung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- the University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Result] Ho FY, Chung KF, Yeung WF, Ng TH, Cheng SK. Weekly brief phone support in self-help cognitive behavioral therapy for insomnia disorder: Relevance to adherence and efficacy. Behav Res Ther. 2014 Dec;63:147-56. doi: 10.1016/j.brat.2014.10.002. Epub 2014 Oct 23. PMID 25461790